CLINICAL TRIAL: NCT05905393
Title: The Protective Role of Preoperative Stimulation of the Distal Limb of the Ileostomy Loop With GABA Before Ileostomy Closure
Brief Title: The Protective Role of GABA Stimulation Before Ileostomy Closure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Wei Guo, associate professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KYLL-202212-066-1
Record Dates: First submitted 2023-05-30; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Ileostomy; Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- preoperative stimulation of the efferent loop with GABA before ileostomy closure surgery (Experimental): Preoperative stimulation of the distal limb of the ileostomy loop with GABA was performed during the 5 days prior to surgery every day. During the process and after it, the patient himself registers the appearance of symptoms after each stimulation session: abdominal pain, emission of gas and stool. Sterile Foley catheter No.14 Ch connected to an infusion set was introduced through the defunctioned bowel to allow the slow infusion, for 10-20 minutes, of a solution with 3000 mg of GABA diluted in 100 ml of 0.9% physiological saline. Each preparation was made under sterile conditions and maintaining the cold chain.
  Interventions: Dietary Supplement: preoperative stimulation of the efferent loop with GABA before ileostomy closure surgery
- control group was stimulated without giving any substance (Sham Comparator): Control group was stimulated without giving any substance. During the process and after it, the patient himself registers the appearance of symptoms after each stimulation session: abdominal pain, emission of gas and stool.
  After 5 stimulation sessions, reconstructive surgery was performed within the following 24 h.
  Interventions: Dietary Supplement: preoperative stimulation of the efferent loop with only physiological saline

INTERVENTIONS:
Dietary Supplement: preoperative stimulation of the efferent loop with GABA before ileostomy closure surgery — Foley catheter No.14 Ch connected to an infusion set was introduced through the defunctioned bowel to allow the slow infusion, for 10-20 minutes, of a solution with 3000 mg of GABA diluted in 100 ml of 0.9% physiological saline.
  Arms: preoperative stimulation of the efferent loop with GABA before ileostomy closure surgery
Dietary Supplement: preoperative stimulation of the efferent loop with only physiological saline — Foley catheter No.14 Ch connected to an infusion set was introduced through the defunctioned bowel to allow the slow infusion, for 10-20 minutes, of 100 ml of 0.9% physiological saline.
  Arms: control group was stimulated without giving any substance

SUMMARY:
The goal of this clinical trial is to explore whether preoperative stimulation of the distal limb of the ileostomy loop with gamma aminobutyric acid (GABA) could effectively reduce the incidence of complications after ileostomy closure.

Participants will be divided into two groups. One group included patients treated with stimulation of the efferent loop with GABA prior to transit reconstruction surgery; the other control group was stimulated without giving any substance.

Researchers will compare incidence of complications such as postoperative ileus, diarrhea and other parameters such as time to tolerating a diet, start of the passage of flatus, start of the passage of stool, postoperative stay, etc.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age;
* body mass index (BMI) 18.5-28 kg/m2;
* having protective ileostomy after colorectal carcinoma surgery free of disease;
* with endoscopic and histological confirmation of diversion colitis;
* no oral antibiotics within 3 months;
* having signed the informed consent.

Exclusion Criteria:

* under 18 years of age;
* clinical history, and histological confirmation of inflammatory bowel disease with colorectal involvement;
* history of neoadjuvant or adjuvant chemoradiotherapy;
* other serious chronic diseases, such as cardiovascular and cerebrovascular diseases, diabetes, respiratory diseases, etc;
* serious perioperative complications such as anastomotic rupture after surgery;
* oral antibiotics within three months;
* participation in any other studies within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
incidence of complications after ileostomy closure | From date of randomization until the date of discharge, assessed up to 20 days
  postoperative ileus, diarrhea, time to tolerating a diet, start of the passage of flatus, start of the passage of stool, postoperative stay.

SECONDARY OUTCOMES:
glucose metabolism-related parameters | From date of randomization until the date of discharge, assessed up to 20 days
  Insulin, C peptide
microbiota alteration | From date of randomization until the date of discharge, assessed up to 20 days
  microbiota alteration before and after GABA stimulation
metabolite alteration | From date of randomization until the date of discharge, assessed up to 20 days
  metabolite alteration before and after GABA stimulation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Strandwitz P, Kim KH, Terekhova D, Liu JK, Sharma A, Levering J, McDonald D, Dietrich D, Ramadhar TR, Lekbua A, Mroue N, Liston C, Stewart EJ, Dubin MJ, Zengler K, Knight R, Gilbert JA, Clardy J, Lewis K. GABA-modulating bacteria of the human gut microbiota. Nat Microbiol. 2019 Mar;4(3):396-403. doi: 10.1038/s41564-018-0307-3. Epub 2018 Dec 10. PMID 30531975
- [Background] Rodriguez-Padilla A, Morales-Martin G, Perez-Quintero R, Gomez-Salgado J, Balongo-Garcia R, Ruiz-Frutos C. Postoperative Ileus after Stimulation with Probiotics before Ileostomy Closure. Nutrients. 2021 Feb 15;13(2):626. doi: 10.3390/nu13020626. PMID 33671968
- [Background] Bansal P, Wang S, Liu S, Xiang YY, Lu WY, Wang Q. GABA coordinates with insulin in regulating secretory function in pancreatic INS-1 beta-cells. PLoS One. 2011;6(10):e26225. doi: 10.1371/journal.pone.0026225. Epub 2011 Oct 21. PMID 22031825
- [Background] Soltani N, Qiu H, Aleksic M, Glinka Y, Zhao F, Liu R, Li Y, Zhang N, Chakrabarti R, Ng T, Jin T, Zhang H, Lu WY, Feng ZP, Prud'homme GJ, Wang Q. GABA exerts protective and regenerative effects on islet beta cells and reverses diabetes. Proc Natl Acad Sci U S A. 2011 Jul 12;108(28):11692-7. doi: 10.1073/pnas.1102715108. Epub 2011 Jun 27. PMID 21709230
- [Background] Garfinkle R, Savage P, Boutros M, Landry T, Reynier P, Morin N, Vasilevsky CA, Filion KB. Incidence and predictors of postoperative ileus after loop ileostomy closure: a systematic review and meta-analysis. Surg Endosc. 2019 Aug;33(8):2430-2443. doi: 10.1007/s00464-019-06794-y. Epub 2019 Apr 17. PMID 31020433
- [Background] Matthiessen P, Hallbook O, Rutegard J, Simert G, Sjodahl R. Defunctioning stoma reduces symptomatic anastomotic leakage after low anterior resection of the rectum for cancer: a randomized multicenter trial. Ann Surg. 2007 Aug;246(2):207-14. doi: 10.1097/SLA.0b013e3180603024. PMID 17667498
- [Background] Wang S, Xiang YY, Zhu J, Yi F, Li J, Liu C, Lu WY. Protective roles of hepatic GABA signaling in acute liver injury of rats. Am J Physiol Gastrointest Liver Physiol. 2017 Mar 1;312(3):G208-G218. doi: 10.1152/ajpgi.00344.2016. Epub 2016 Dec 15. PMID 27979827
- [Background] Wang S, Sui S, Liu Z, Peng C, Liu J, Luo D, Fan X, Liu C, Lu WY. Protective roles of hepatic gamma-aminobutyric acid signaling in acute ethanol exposure-induced liver injury. J Appl Toxicol. 2018 Mar;38(3):341-350. doi: 10.1002/jat.3544. Epub 2017 Oct 17. PMID 29044621
- [Background] Beamish EL, Johnson J, Shaw EJ, Scott NA, Bhowmick A, Rigby RJ. Loop ileostomy-mediated fecal stream diversion is associated with microbial dysbiosis. Gut Microbes. 2017 Sep 3;8(5):467-478. doi: 10.1080/19490976.2017.1339003. Epub 2017 Jun 16. PMID 28622070
- [Background] Rombey T, Panagiotopoulou IG, Hind D, Fearnhead NS. Preoperative bowel stimulation prior to ileostomy closure to restore bowel function more quickly and improve postoperative outcomes: a systematic review. Colorectal Dis. 2019 Sep;21(9):994-1003. doi: 10.1111/codi.14636. Epub 2019 May 7. PMID 30963659